CLINICAL TRIAL: NCT02963402
Title: Analysis of Immunoregulatory Mechanisms of Treg Cells Induced by Tocilizumab
Brief Title: Immunoregulatory Mechanisms of Treg Cells Induced by Tocilizumab
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TOC-2016-09
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Arthritis,Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tocilizumab treated
  Interventions: Drug: Tocilizumab
- Anti-TNF treated
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Tocilizumab
  Groups: Tocilizumab treated
Drug: Adalimumab
  Groups: Anti-TNF treated

SUMMARY:
We can speculate that the best responders to tocilizumab should have multiple related elements (Treg CD39, adenosine, IL-35) successfully induced and expressed in order to play its beneficial role. The study of these elements and its pathways could help identify the best responders to tocilizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all sexes, aged ≥ 18 years.
* RA Patients (according to ACR / EULAR criteria 2010) of moderate to severe activity (DAS 28> 3.2 or SDAI> 11), and 6 months or more of evolution, starting treatment with ACTEMRA (tocilizumab) or with an anti-TNF, according to the product data.
* Patients with body weight ≤ 150 kg.
* Patients who have received written information about the study and gave their informed consent to participate in the study

Exclusion Criteria:

* Patients with a history of autoimmune disease or inflammatory joint disease other than RA.
* Patients treated with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is greater) before starting treatment with tocilizumab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AR patients treated with tocilizumab in monotherapy or treated with adalimumab as control.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Treg phenotype | Baseline to 6 months change
ATP (adenosine triphosphate) | Baseline to 6 months change

CONTACTS AND LOCATIONS:
Locations (1):
- Insitut de Recerca Hospital de la Santa Creu i Sant Pau, Barcelona, Spain